CLINICAL TRIAL: NCT02185209
Title: Surgical Treatment of Peri-implantitis With and Without Systemically Adjunctive Antibiotics A Prospective, Double Blind, Randomized, Three Armed, Parallel, Placebo Controlled Clinical Trial
Brief Title: Surgical Treatment of Peri-implantitis With and Without Systemically Adjunctive Antibiotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Margareta Hultin (Other)
Responsible Party: Sponsor-Investigator, Margareta Hultin, DDS, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PERI-IMPL
Record Dates: First submitted 2014-06-23; First posted 2014-07-09 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Periodontal Diseases; Periimplantitis
MeSH Terms: conditions — Periodontal Diseases; Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Experimental): Patients with periimplantitis undergoing surgical treatment with will receive placebo three times daily (TID)
  Interventions: Drug: Placebo
- amoxicillin + metronidazole (Active Comparator): Patients with periimplantitis undergoing surgical treatment with amoxicillin (500 mg TID) + metronidazole (400 mg TID) for 7 days
  Interventions: Drug: Amoxicillin Sandoz; Drug: Metronidazole Sanofi
- phenoxymetylpencillin + metronidazol (Active Comparator): Patients with periimplantitis undergoing surgical treatment with phenoxymetylpencillin, (800mg×2 TID) + metronidazol (400 mg TID) for 7 days
  Interventions: Drug: Metronidazole Sanofi; Drug: Phenoxymethylpenicillin Meda

INTERVENTIONS:
Drug: Placebo — Place capsule to mimic antibiotics
  Arms: Placebo
Drug: Amoxicillin Sandoz — Tablet 500 mg amoxicillin Sandoz three times a day
  Arms: amoxicillin + metronidazole
Drug: Metronidazole Sanofi — 400 mg metronidazole Sanofi administered three times a day (TID)
  Arms: amoxicillin + metronidazole; phenoxymetylpencillin + metronidazol
Drug: Phenoxymethylpenicillin Meda — 1600 mg phenoxymethylpenicillin Meda, three time a day (TID)
  Arms: phenoxymetylpencillin + metronidazol

SUMMARY:
The purpose of this study is to investigate if the use of systemic adjunctive antibiotics in the treatment of periimplantitis is needed.

DETAILED DESCRIPTION:
This study will give the opportunity to draw scientifically based conclusions on the recommendations of the use of adjunctive systemic antibiotics in the treatment of peri-implantitis. This study will also be able to determine the ecological impact on the oropharyngeal and intestinal microflora between different antibiotic treatments. The lack of knowledge in this area has been highlighted by the Food and Drug Administration and The Swedish Council on Health Technology Assessment (SBU)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18-65 year
2. Patients who has been referred by a general dentist to a specialist clinic in periodontology for treatment of peri-implantitis.
3. Having sign of peri-implantitis around at least one osseointegrated dental implant that has been in function for ≥ one year
4. Peri-implantitis is diagnosed when; PPD of ≥ 6mm can be found at a dental implant in association with BOP and/or suppuration together with the loss of marginal alveolar bone of more than 2 mm detected on intraoral radiographs (giving radiographic exposure of at least ≥ 3 fixture threads).
5. Partially or completely edentulous subjects with healthy or treated periodontal conditions enrolled in a regular supportive program.
6. Full-Mouth Plaque Score (FMPS) ≤ 25
7. Signed informed consent

Exclusion Criteria:

1. Known allergy to amoxicillin, penicillin (PcV), metronidazole or betalactamic
2. Contraindication for dental surgical treatment (i.e. immunocompromised, uncontrolled DM (B-GHb-A1C 8-9 %, 64-75 mmol/mol), osteoporosis, I.V bisphosphonate treatment due to malignancy, pregnant and lactating women).
3. Incapability to perform basal oral hygiene measures due to physical or mental disorders.
4. Received systemic antimicrobial therapy in the past three months.
5. Currently on allopurinol, digoxin, disulfiram, lithium, busulfan, 5-fluorouracil, methotrexate, phenytoin, cyclosporine and warfarin.
6. Known severe chronic peripheral or central disease of the nervous system
7. Known alcohol abuse
8. Known hepatic encephalopathy
9. Known lactose intolerance, galactose intolerance
10. Untreated periodontal condition.
11. Implant showing sign of mobility.
12. Implants with bone loss exceeding 2/3 of the length of the implant or implants with bone loss beyond any transverse openings in hollow implants.
13. Any medical condition or on any concomitant medication that, in the opinion of the investigator, might interfere with the evaluation of the study objectives or jeopardize patient safety

Patients with xerostomia or having slow bowel motion will be excluded from the group of patients providing salivary and fecal samples.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-03; Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth change and bone level stability | 0,6 and 12 months

SECONDARY OUTCOMES:
Change of clinical soft tissue inflammation, bleeding on probing (BOP) | 0, post operative 12 month
Soft tissue recession (REC) and clinical attachment level gain (CAL) | 0,6 and 12 month
• Quantitative and qualitative change in levels of the peri-implant periopathogenic microflora | 0,6 and 12 months
• Susceptibility changes of the oral and intestinal microflora to amoxicillin, metronidazole and penicillin. | 0,6 and 12 month
Quantitative and qualitative changes in the oral and intestinal microflora | 0,6 and 12 month
Concentration of amoxicillin, metronidazole and PcV in saliva and feces | 0, 6 and 12 month
• Follow-up of adverse events related or unrelated to the investigated medical products | 0,6, and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Hultin, DDSass. prof, Study Chair — Karolinska Institute, Dental medicine; Bodil Lund, DDSass.prof, Study Director — Karolinska Institute, Dental Medicine; Dalia Kahlil, DDS, PhDstud, Principal Investigator — Karolinska Institute, Dental Medicine
Locations (2):
- Sweden (2):
  - Folktandvården Skanstull, Stockholm
  - Folktandvården Kaniken, Uppsala

REFERENCES:
- [Derived] Riben Grundstrom C, Lund B, Kampe J, Belibasakis GN, Hultin M. Systemic antibiotics in the surgical treatment of peri-implantitis: A randomized placebo-controlled trial. J Clin Periodontol. 2024 Aug;51(8):981-996. doi: 10.1111/jcpe.13994. Epub 2024 May 3. PMID 38699828